CLINICAL TRIAL: NCT02313103
Title: Single-dose Pharmacokinetics and Safety of Oral Lofexidine in Renally-Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USWM-LX1-1008; 1R01DA030916 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Renally Impaired Subjects
Keywords: ESRD; End Stage Renal Disease; Normal Healthy Volunteers; Renally Impaired
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lofexidine HCl (Other): End Stage Renal Disease (ESRD) subjects will be dosed with 400 micrograms of lofexidine HCl with 240 mL water after their hemodialysis session.
  Interventions: Drug: lofexidine HCl
- Matched Control (Other): normal renal function subjects (enrolled to match each End Stage Renal Disease subject) will be dosed with 400 micrograms of lofexidine HCl with 240 mL water at the same clock time as ESRD subjects.
  Interventions: Drug: lofexidine HCl

INTERVENTIONS:
Drug: lofexidine HCl — 400 micrograms

SUMMARY:
This is a phase 1, open-label, parallel-group, single-dose study of lofexidine in 8 adult subjects with ESRD maintained on hemodialysis (3 times per week) and 8 control subjects with normal renal function, recruited as 1:1 matches to each ESRD subjects, matched for gender, age, and BMI.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, parallel-group, single-dose study of lofexidine in 8 adult subjects with ESRD maintained on hemodialysis (3 times per week) and 8 control subjects with normal renal function (creatinine [Cr] clearance >90 mL/min), recruited as 1:1 matches to each ESRD subject, matched for gender, age (±10 years), and body mass index (BMI) (±15%). Normal renal function and ESRD subjects will be confined to an inpatient facility from the day before dosing to 144 or 156 hours after dosing, respectively, for a total of 7 8 nights and 8-9 days of inpatient confinement.

Subjects who successfully complete screening will report to the inpatient facility at an appropriate time the day before study drug administration to undergo pre-dosing study procedures (Day 1). The next morning (Day 1), all subjects will receive breakfast (approximately 6 hours before planned lofexidine dosing) and then ESRD subjects will begin their hemodialysis session. All subjects will receive a single, oral dose of 400 µg lofexidine HCl (two 200 µg tablets), dosed with 240 mL of water, the clock time for which will be approximately the same for both normal renal function subjects and ESRD subjects. Because ESRD subjects will be maintained on 3 times per week dialysis, lofexidine will be administered near the beginning of a 3-day between-dialysis interval.

Fingerprick blood samples for subjects with normal renal function will be collected for PK analysis at multiple time points over the next 144 hours. Fingerprick blood samples for ESRD subjects will be collected for PK analysis at multiple time points over the next 156 hours. Fingerprick blood samples (0.5 mL each) will be collected in BD Microtainer pink top K2EDTA tubes.

Two (2) venous blood samples (4-6 mL each in K2EDTA tubes) will be collected from each subject for lofexidine protein binding analysis, one sample collected 0-60 minutes before dosing and one sample collected 4 hours post-dose.

Pooled urine samples for subjects with normal renal function will be collected at 0 3 hours, 3 6 hours, 6 12 hours, 12 24 hours, 24 48 hours, 48 72 hours, 72 96 hours, and 96 144 hours post-dose. Pooled urine samples will be collected from ESRD subjects as available according to the same schedule.

Arterial and venous blood samples from the arterial-venous (A-V) shunt (0.5 mL in BD Microtainer pink top K2EDTA tubes) for PK analysis will be collected from ESRD subjects at 0.5, 1.5, 2.5, and 3.5 hours into each of the two 4 hour hemodialysis sessions. Additionally, fingerprick blood samples (0.5 mL) will be collected from the hand contralateral to the arm used for the dialysis A V shunt at each of these specified time points. Dialysate from ESRD subjects will be collected during the two 4 hour hemodialysis sessions at 0 1 hour, 1 2 hour, 2 3 hour, and 3 4 hour. Two 10 mL samples from each of the 1-hour pooled dialysate collections will be aliquoted into suitable collection tubes.

Safety will be assessed by recording adverse events (AEs), measuring vital signs (blood pressure and pulse rate) and clinical laboratory tests (chemistry, hematology, and urinalysis), recording 12 lead safety and Holter electrocardiograms (ECGs), and performing physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-75 years at enrollment with a BMI between 18 and 38 kg/m2, inclusive. Subjects with normal renal function: gender, age (±10 years), and BMI (±15%) matched to their ESRD subject.
* Male or female; however, if female: must be using contraception if of childbearing potential or must be surgically sterile; and must not be lactating.
* Subjects with ESRD must have been receiving adequate maintenance hemodialysis (at least 3 times per week) for at least 3 months before Day -1 (i.e., approximate Kt/V >1.1 based on subject's nephrologist and Investigator); subjects with normal renal function must have a creatinine clearance (CLcr) of less than or equal to 90 mL/min as estimated by Cockcroft and Gault or, if clinically indicated, by a 24 hour urine CLcr test.
* Subjects with ESRD must be on a stable medication program, except for medications prescribed for maintenance of hemoglobin, for at least 2 weeks before Day 1.
* At screening a matched control subject is in good health based on medical history, physical exam, laboratory profile, and ECG as judged by the Investigator.
* If subject smokes, subject agrees to limit smoking while in the study to not more than 10 cigarettes per day.
* Provides written informed consent before participation in the study, and an appropriate HIPAA (Health Insurance Portability and Accountability Act) form is signed and dated.

Exclusion Criteria:

* Fails to meet all of the inclusion criteria.
* The matched control subject has a history of clinically significant disease, including cardiovascular, gastrointestinal (GI), renal, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease or the ESRD subject has a history of clinically significant disease including cardiovascular, GI, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, or collagen disease.
* Females: pregnant, breastfeeding, planning to become pregnant, or a positive pregnancy test.
* Clinically significant illness other than renal disease or known conditions associated with renal disease for ESRD subjects, within 4 weeks before Day -1.
* Use of herbal supplements within 3 weeks before Day 1.
* Received treatment of more than a single dose of CYP3A4 inducer (e.g., rifampin, barbiturates, phenytoin, glucocorticoids, St. John's Wort) within 4 weeks before Day -1.
* Received treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, diltiazem, macrolides antibiotics) within 2 weeks before Day -1.
* Currently taking any medication identified as potentially producing QTc prolongations of 10 msec or greater.
* Received an investigational medication during the last month (30 days) preceding Day -1.
* Consumes more than 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) or has a significant history of alcohol abuse or drug/chemical abuse within the last 1 year.
* Consumed grapefruit or grapefruit juice within 4 days before Day 1.
* Positive urine or saliva (ESRD subjects) drug screen and alcohol breathalyzer test, unless positive result is due to an approved prescribed medication (pain medication or benzodiazepine).
* Positive human immunodeficiency virus (HIV) test or tests positive for hepatitis B surface antigen.
* Known allergy or intolerance to any compound in the test product or any other closely related compound.
* Donated blood/plasma exceeding 500 mL, during the 3 month period before Day 1.
* Abnormal electrolyte values, including any including any pre-dialysis values in ESRD subjects outside of the following ranges: potassium 3.0-6.5 mmol/L; calcium 7.0-11.0 mg/dL; sodium: 120 150 mmol/L.
* Abnormal cardiovascular exam at Screening, including any of the following: clinically significant abnormal ECG at Screening (e.g., second or third degree heart block, uncontrolled arrhythmia, QTcF [Fridericia's correction] interval >450 msec for males and >470 msec for females); heart rate <45 bpm or symptomatic bradycardia; systolic blood pressure <90 mmHg or symptomatic hypotension; blood pressure >180/105 mmHg; or prior history of myocardial infarction within 1 year before Day 1.
* Subjects with normal renal function will not be eligible to participate in the study if any of the following exclusion criteria also apply: Received any over-the-counter medication, including topical medications, vitamins, and nutritional supplements or any prescription medication (except female hormonal contraceptives or hormone replacement therapy) within 14 days or 5 half lives (whichever is less) before Day 1.
* Subjects with ESRD will not be eligible to participate in the study if any of the following exclusion criteria also apply: Recipient of a functioning transplanted solid organ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PK Profile | pre dose until 156 hours post dose
  Cmax, Tmax, AUC, λz, CL/F, T½, CLr, CLd, Ae

SECONDARY OUTCOMES:
Adverse events | screening through day 7 or 8
Clinical laboratory tests | screening through day 7 or 8
  hematology, chemistry and urinalysis
Vital signs | screening through day 7 or 8
  blood pressure and pulse
12-lead ECG | screening through day 7 or 8
holter ECG | screening through day 7 or 8

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — OCRS; James Longstreth, PhD, Study Director — USWM, LLC (dba US WorldMeds); Charles Gorodetzky, MD, Study Director — USWM, LLC (dba US WorldMeds)
Locations (1):
- Orlando, Florida, United States